CLINICAL TRIAL: NCT00919633
Title: COPE-HCV: Continuous Interferon Delivery Via the Medtronic Paradigm Pump Infusion System Clinical Evaluation for Chronic HCV
Brief Title: Safety and Efficacy Study to Compare Continuous Infusion of Interferon With Standard of Care for Chronic Hepatitis C
Acronym: COPE-HCV
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Medtronic Corporate Technologies and New Ventures (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 4316001
Record Dates: First submitted 2009-06-10; First posted 2009-06-12 (Estimated); Results first posted 2014-04-30 (Estimated); Last update posted 2019-10-09 (Actual); Status verified 2019-09

CONDITIONS: Hepatitis C
Keywords: hepatitis C; HCV; genotype; sustained virological response; rapid virological response; interferon
MeSH Terms: conditions — Hepatitis C | interventions — Interferon alpha-2; peginterferon alfa-2b; Ribavirin

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Group 1: interferon alfa-2b (dose 1) (Experimental): continuous subcutaneous infusion for 48 weeks
  Interventions: Drug: interferon alfa-2b; Drug: ribavirin, USP; Device: external drug infusion pump
- Group 2: interferon alfa-2b (dose 2) (Experimental): continuous subcutaneous infusion for 48 weeks
  Interventions: Drug: interferon alfa-2b; Drug: ribavirin, USP; Device: external drug infusion pump
- Group 3: interferon alfa-2b (dose 3) (Experimental): continuous subcutaneous infusion for 48 weeks
  Interventions: Drug: interferon alfa-2b; Drug: ribavirin, USP; Device: external drug infusion pump
- Group 4: peginterferon alfa-2b (1.5 μg/kg) (Active Comparator): subcutaneous weekly for 48 weeks
  Interventions: Drug: peginterferon alfa-2b; Drug: ribavirin, USP

INTERVENTIONS:
Drug: interferon alfa-2b — subcutaneous continuous infusion at one of three doses for 48 weeks
  Other Names: INTRON® A
  Arms: Group 1: interferon alfa-2b (dose 1); Group 2: interferon alfa-2b (dose 2); Group 3: interferon alfa-2b (dose 3)
Drug: peginterferon alfa-2b — 1.5 μg/kg subcutaneous weekly for 48 weeks
  Other Names: PEGINTRON™
  Arms: Group 4: peginterferon alfa-2b (1.5 μg/kg)
Drug: ribavirin, USP — All patients will receive oral ribavirin
  Other Names: Rebetol®
Device: external drug infusion pump — pump delivery system for continuous subcutaneous infusion of interferon alfa-2b
  Other Names: Medtronic MiniMed™ Paradigm® Insulin Pump Infusion System
  Arms: Group 1: interferon alfa-2b (dose 1); Group 2: interferon alfa-2b (dose 2); Group 3: interferon alfa-2b (dose 3)

SUMMARY:
The purpose of the study is to evaluate if continuous subcutaneous delivery of interferon alfa-2b using an external drug pump in combination with the use of oral ribavirin provides a safe and effective treatment for patients with chronic hepatitis C infection as compared to patients who receive standard treatment.

DETAILED DESCRIPTION:
The study will include patients who are diagnosed with chronic hepatitis C genotype 1 infection and who have received no previous interferon or other anti-HCV treatment.

ELIGIBILITY:
Inclusion Criteria:

* Signed patient consent form
* Genotype 1 chronic HCV with detectable HCV RNA
* No previous treatment for HCV infection
* Hepatitis B and human immunodeficiency virus negative at screening visit
* Able and willing to follow contraception requirements
* Screening laboratory values, test, and physical exam within acceptable ranges
* Weight between 40 kg and 125 kg
* Proficiency in the use of the external pump infusion system

Exclusion Criteria:

* Current or planned enrollment in another investigational device or drug study
* Anticipated inability to complete all clinic visits and comply with study procedures
* History of, or any current medical condition, which could impact the safety of the subject during the study
* Autoimmune hepatitis, suspected hepatocellular carcinoma, decompensated liver disease, or other known liver disease other than HCV
* Alcoholism or substance abuse with <6 documented months of sobriety
* Known allergy or sensitivity to interferons or ribavirin
* Any other condition that, in the opinion of the Investigator, would make the subject unsuitable for enrollment or could interfere with the subject participating in and completing the study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 116 (Actual)
Dates: Start 2009-06; Primary Completion 2012-07 (Actual); Study Completion 2012-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Muir, M.D., Principal Investigator — Duke Clinical Research Institute; Sarah Mische, PhD, Study Director — Medtronic Ventures and New Therapies
Locations (1):
- Duke Clinical Research Institute, Durham, North Carolina, United States

REFERENCES:
- See also: Common terminology criteria for adverse events, version 3.0 — http://ctep.cancer.gov
- See also: International Committee of Medical Journal Editors. Uniform requirements for manuscripts submitted to biomedical journals: writing and editing for biomedical publication. Publication ethics: sponsorship, authorship and accountability. — http://www.ICMJE.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Enrollment 09-Jun-2009, final subject complete 19-Jun-2012.
Pre-assignment Details: 210 screened, 116 randomized, 106 received at least 1 dose of study drug.
Groups:
- Group 4: Peginterferon Alfa-2b (1.5 μg/kg): subcutaneous weekly for 48 weeks
  peginterferon alfa-2b : 1.5 μg/kg subcutaneous weekly for 48 weeks
  ribavirin, USP : All patients will receive oral ribavirin
- Group 1: Interferon Alfa-2b (Dose 1); Group 2: Interferon Alfa-2b (Dose 2); Group 3: Interferon Alfa-2b (Dose 3): continuous subcutaneous infusion for 48 weeks
  external drug infusion pump : pump delivery system for continuous subcutaneous infusion of interferon alfa-2b
  interferon alfa-2b : subcutaneous continuous infusion at one of three doses for 48 weeks
  ribavirin, USP : All patients will receive oral ribavirin
Period: Overall Study
Arm/Group | Group 4: Peginterferon Alfa-2b (1.5 μg/kg) | Group 1: Interferon Alfa-2b (Dose 1) | Group 2: Interferon Alfa-2b (Dose 2) | Group 3: Interferon Alfa-2b (Dose 3)
Started | 28 | 25 | 27 | 26
Completed | 6 | 10 | 4 | 5
Not Completed | 22 | 15 | 23 | 21
Not completed — Adverse Event | 1 | 9 | 12 | 10
Not completed — Death | 0 | 0 | 2 | 0
Not completed — Lack of Efficacy | 17 | 3 | 2 | 3
Not completed — Withdrawal by Subject | 1 | 2 | 4 | 3
Not completed — Lost to Follow-up | 3 | 1 | 0 | 2
Not completed — Withdraw consent post transition to SOC | 0 | 0 | 1 | 1
Not completed — Protocol Violation | 0 | 0 | 0 | 1
Not completed — Physician Decision | 0 | 0 | 0 | 1
Not completed — Request of withdrawal w/o future contact | 0 | 0 | 1 | 0
Not completed — Viral rebound outside protocol timepoint | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Group 4: Peginterferon Alfa-2b (1.5 μg/kg) | Group 1: Interferon Alfa-2b (Dose 1) | Group 2: Interferon Alfa-2b (Dose 2) | Group 3: Interferon Alfa-2b (Dose 3) | Total
Number analyzed (Participants) | 28 | 25 | 27 | 26 | 106
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 28 | 25 | 27 | 26 | 106
  >=65 years | 0 | 0 | 0 | 0 | 0
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 51.2 [48.5 to 53.8] | 51.5 [47.0 to 56.1] | 51.3 [46.7 to 55.5] | 49.1 [44.6 to 53.2] | 51.2 [44.6 to 56.1]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 12 | 11 | 12 | 43
  Male | 20 | 13 | 16 | 14 | 63
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 3 | 3 | 4 | 12
  Not Hispanic or Latino | 26 | 22 | 24 | 22 | 94
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 0 | 1 | 2
  Asian | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 1 | 0 | 1
  Black or African American | 5 | 2 | 4 | 3 | 14
  White | 21 | 23 | 22 | 21 | 87
  More than one race | 1 | 0 | 0 | 1 | 2
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 28 | 25 | 27 | 26 | 106
Hepatitis C Genotype [Number; unit: participants] — 1a, 1b
  participants
    1a | 24 | 19 | 23 | 19 | 85
    1b | 4 | 6 | 4 | 7 | 21

OUTCOME MEASURES:

1. Primary Outcome: Viral Load: Incidence of Sustained Virologic Response (SVR)
Time Frame: 24 weeks after treatment is complete
Measure: Number; unit: participants
Arm/Group | Group 4: Peginterferon Alfa-2b (1.5 μg/kg) | Group 1: Interferon Alfa-2b (Dose 1) | Group 2: Interferon Alfa-2b (Dose 2) | Group 3: Interferon Alfa-2b (Dose 3)
Number analyzed (Participants) | 28 | 25 | 27 | 26
participants | 4 | 7 | 2 | 4

2. Secondary Outcome: Rapid Virologic Response (RVR)
Time Frame: Study Week 4
Measure: Number; unit: participants
Arm/Group | Group 4: Peginterferon Alfa-2b (1.5 μg/kg) | Group 1: Interferon Alfa-2b (Dose 1) | Group 2: Interferon Alfa-2b (Dose 2) | Group 3: Interferon Alfa-2b (Dose 3)
Number analyzed (Participants) | 28 | 25 | 27 | 26
participants | 2 | 4 | 7 | 11

3. Secondary Outcome: Early Virologic Response (EVR)
Time Frame: Study week 12
Measure: Number; unit: participants
Arm/Group | Group 4: Peginterferon Alfa-2b (1.5 μg/kg) | Group 1: Interferon Alfa-2b (Dose 1) | Group 2: Interferon Alfa-2b (Dose 2) | Group 3: Interferon Alfa-2b (Dose 3)
Number analyzed (Participants) | 28 | 25 | 27 | 26
participants | 7 | 15 | 13 | 11

ADVERSE EVENTS:
Time Frame: Adverse events were collected the duration of the study from activation to closure.
Groups:
- PEGINTRON 1.5: subcutaneous weekly for 48 weeks
  peginterferon alfa-2b : 1.5 μg/kg subcutaneous weekly for 48 weeks
  ribavirin, USP : All patients will receive oral ribavirin
- INTRON A 80,000; INTRON A 120,000; INTRON A 160,000: continuous subcutaneous infusion for 48 weeks
  external drug infusion pump : pump delivery system for continuous subcutaneous infusion of interferon alfa-2b
  interferon alfa-2b : subcutaneous continuous infusion at one of three doses for 48 weeks
  ribavirin, USP : All patients will receive oral ribavirin
Arm/Group | PEGINTRON 1.5 | INTRON A 80,000 | INTRON A 120,000 | INTRON A 160,000
Serious Adverse Events (participants affected / at risk) | 2/28 | 6/25 | 5/27 | 6/26
Other Adverse Events (participants affected / at risk) | 28/28 | 25/25 | 27/27 | 26/26
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | PEGINTRON 1.5 (N=28) | INTRON A 80,000 (N=25) | INTRON A 120,000 (N=27) | INTRON A 160,000 (N=26)
Bronchitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cellulitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Injection Site Cellulitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Staphylococcal Abscess (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Appendicitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 2 (2) | 2 (2) | 0 (0)
Pneumonia Moraxella (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Streptococcal Abscess (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Melaena (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Musculoskeletal Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Musculoskeletal Chest Pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Suicidal Ideation (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Suicide Attempt (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Arteriosclerosis Coronary Artery (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypertensive Heart Disease (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Liver Disorder (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Type 2 Diabetes Mellitus (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | PEGINTRON 1.5 (N=28) | INTRON A 80,000 (N=25) | INTRON A 120,000 (N=27) | INTRON A 160,000 (N=26)
Fatigue (General disorders) | 14 (14) | 16 (16) | 15 (15) | 16 (16)
Influenza Like Illness (General disorders) | 11 (11) | 8 (8) | 9 (9) | 11 (11)
Pyrexia (General disorders) | 7 (7) | 10 (10) | 11 (11) | 9 (9)
Asthenia (General disorders) | 0 (0) | 0 (0) | 3 (3) | 5 (5)
Chills (General disorders) | 10 (10) | 6 (6) | 3 (3) | 5 (5)
Irritability (General disorders) | 4 (4) | 5 (5) | 5 (5) | 5 (5)
Oedema Peripheral (General disorders) | 0 (0) | 0 (0) | 2 (2) | 3 (3)
Non-Cardiac Chest Pain (General disorders) | 0 (0) | 2 (2) | 1 (1) | 2 (2)
Pain (General disorders) | 9 (9) | 4 (4) | 2 (2) | 2 (2)
Nausea (Gastrointestinal disorders) | 10 (10) | 15 (15) | 13 (13) | 18 (18)
Vomiting (Gastrointestinal disorders) | 1 (1) | 2 (2) | 6 (6) | 8 (8)
Diarrhoea (Gastrointestinal disorders) | 4 (4) | 4 (4) | 8 (8) | 6 (6)
Constipation (Gastrointestinal disorders) | 1 (1) | 1 (1) | 3 (3) | 3 (3)
Dry Mouth (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2) | 2 (2)
Stomatitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 3 (3) | 2 (2)
Abdominal Pain (Gastrointestinal disorders) | 0 (0) | 2 (2) | 3 (3) | 1 (1)
Abdominal Pain Upper (Gastrointestinal disorders) | 1 (1) | 0 (0) | 2 (2) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 2 (2) | 1 (1)
Gingival Pain (Gastrointestinal disorders) | 1 (1) | 0 (0) | 2 (2) | 0 (0)
Headache (Nervous system disorders) | 11 (11) | 15 (15) | 18 (18) | 17 (17)
Dizziness (Nervous system disorders) | 1 (1) | 6 (6) | 9 (9) | 4 (4)
Disturbance in Attention (Nervous system disorders) | 0 (0) | 2 (2) | 3 (3) | 3 (3)
Memory Impairment (Nervous system disorders) | 1 (1) | 2 (2) | 3 (3) | 2 (2)
Dysgeusia (Nervous system disorders) | 1 (1) | 1 (1) | 4 (4) | 0 (0)
Hypersomnia (Nervous system disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Hypogeusia (Nervous system disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 9 (9) | 7 (7) | 7 (7) | 11 (11)
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 (3) | 1 (1) | 6 (6) | 6 (6)
Back Pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2) | 5 (5) | 5 (5)
Muscle Spasms (Musculoskeletal and connective tissue disorders) | 2 (2) | 6 (6) | 4 (4) | 2 (2)
Muscular Weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
Cellulitis (Infections and infestations) | 2 (2) | 0 (0) | 2 (2) | 3 (3)
Upper Respiratory Tract Infection (Infections and infestations) | 2 (2) | 5 (5) | 5 (5) | 3 (3)
Bronchitis (Infections and infestations) | 0 (0) | 4 (4) | 4 (4) | 0 (0)
Urinary Tract Infection (Infections and infestations) | 1 (1) | 0 (0) | 2 (2) | 1 (1)
Sinusitis (Infections and infestations) | 1 (1) | 2 (2) | 2 (2) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 8 (8) | 4 (4) | 7 (7)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 4 (4) | 8 (8) | 6 (6)
Productive Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2) | 3 (3) | 3 (3)
Oropharyngeal Pain (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (2) | 1 (1) | 2 (2)
Respiratory Tract Congestion (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 3 (3) | 4 (4) | 2 (2)
Nasal Congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 2 (2) | 1 (1)
Sinus Congestion (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1) | 2 (2) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 3 (3) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 4 (4) | 5 (5) | 9 (9) | 9 (9)
Anaemia (Blood and lymphatic system disorders) | 7 (7) | 5 (5) | 13 (13) | 4 (4)
Thrombocytopenia (Blood and lymphatic system disorders) | 3 (3) | 5 (5) | 6 (6) | 3 (3)
Leukopenia (Blood and lymphatic system disorders) | 2 (2) | 2 (2) | 2 (2) | 2 (2)
Depression (Psychiatric disorders) | 5 (5) | 11 (11) | 7 (7) | 8 (8)
Insomnia (Psychiatric disorders) | 11 (11) | 6 (6) | 5 (5) | 7 (7)
Anxiety (Psychiatric disorders) | 3 (3) | 4 (4) | 4 (4) | 1 (1)
Confusional State (Psychiatric disorders) | 0 (0) | 2 (2) | 2 (2) | 0 (0)
Libido Decreased (Psychiatric disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Decreased Appetite (Metabolism and nutrition disorders) | 4 (4) | 5 (5) | 8 (8) | 11 (11)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 2 (2) | 0 (0) | 1 (1)
Alopecia (Skin and subcutaneous tissue disorders) | 3 (3) | 10 (10) | 8 (8) | 7 (7)
Rash (Skin and subcutaneous tissue disorders) | 6 (6) | 7 (7) | 6 (6) | 6 (6)
Erythema (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 3 (3)
Pruritus (Skin and subcutaneous tissue disorders) | 4 (4) | 2 (2) | 6 (6) | 3 (3)
Dry Skin (Skin and subcutaneous tissue disorders) | 3 (3) | 4 (4) | 1 (1) | 2 (2)
Dermatitis (Skin and subcutaneous tissue disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Blood Uric Acid Increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Weight Decreased (Investigations) | 1 (1) | 2 (2) | 3 (3) | 2 (2)
Photophobia (Eye disorders) | 0 (0) | 3 (3) | 0 (0) | 1 (1)
Visual Acuity Reduced (Eye disorders) | 0 (0) | 2 (2) | 0 (0) | 1 (1)
Dry Eye (Eye disorders) | 0 (0) | 1 (1) | 2 (2) | 0 (0)
Eye Pain (Eye disorders) | 0 (0) | 1 (1) | 2 (2) | 0 (0)
Retinal Exudates (Eye disorders) | 0 (0) | 2 (2) | 1 (1) | 0 (0)
Angina Pectoris (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Techycardia (Cardiac disorders) | 1 (1) | 3 (3) | 0 (0) | 0 (0)
Ear Pain (Ear and labyrinth disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other